CLINICAL TRIAL: NCT01261260
Title: The Effect of Uridine on GABA and High Energy Phosphate Levels in Healthy Volunteers
Brief Title: Effect of Uridine on GABA and High Energy Phosphate Levels in Healthy Volunteers
Acronym: Uridine-GABA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Perry F. Renshaw MD PhD, Brain Institute, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 2005-P-002083-McLean; 2R01MH058681-04A2 (NIH)
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Healthy Male Subjects
Keywords: uridine; gamma-amino butyric acid; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Proton Echo-Planar Spectroscopic Imaging
MeSH Terms: interventions — Uridine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Uridine (Placebo Comparator): 1g BID
  Interventions: Drug: Uridine

INTERVENTIONS:
Drug: Uridine — 1 gram tablets BID for 7 days

SUMMARY:
On the dual basis of findings indicating GABA increases following acute and eight week SSRI/dopamine agonist administration and those indicating GABA-ergic effects following 14 day pyrimidine administration, the purpose of this study is to assess our following hypotheses:

1. Relative to placebo, an oral dose of 1g of uridine BID for seven days will increase brain GABA levels in a sample of healthy, unmedicated adult males;
2. Relative to placebo, an oral dose of 1g of uridine BID for seven days will increase NTP levels in a sample of healthy, unmedicated adult males; and
3. Brain GABA levels will be directly correlated to high energy phosphate levels in this sample of healthy, unmedicated adult males.

DETAILED DESCRIPTION:
Based on prior MRS studies by our group as well as the work of others, we hypothesize that oral administration of uridine will actuate an increase in brain gamma-amino butyric acid (GABA) levels, along with beta-nucleotide triphosphate (ß-NTP) levels, as compared with baseline. Our aim is to investigate this specific neuropharmacological effect and to demonstrate the suitability of a novel magnetic resonance spectroscopy protocol in so doing. Our rationale includes the consideration that the clinical utility of an intervention demonstrably effective in elevating brain GABA and high energy phosphate levels is broad, since lowered GABA and bioenergetic states are associated with a plurality of affective, anxiety, and substance use disorders.

On the dual basis of findings indicating GABA increases following acute and eight week SSRI/dopamine agonist administration and those noting GABA-ergic effects of 14 day pyrimidine administration, we hypothesize that an oral dose of 2g of uridine per day for seven days will increase brain GABA levels in a sample of healthy, unmedicated adult males. We also hypothesize that this 2g dose of uridine per day for 7 days will increase ß-NTP levels and, further, that the increase in GABA and high energy phosphate levels will be correlated. Of note, the phosphorylation of glutamic acid decarboxylase by ATP significantly increased the activity of this enzyme, which is reponsable for the synthesis of GABA. This choice of time period will allow a determination of time course to efficacy between the acute and extended ranges, and further, because therapeutic dosage levels of uridine have yet to be established, in this and future studies we hope to determine the optimal dosage at which uridine increases brain GABA and ß-NTP levels.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age range of 18-60 years
* BMI between 18.5 and 28
* Medication-free
* Capable of providing informed consent
* Non- smoking for a minimum of one year

Exclusion Criteria:

* Meets DSM-IV criteria for any Axis I disorder (past or present)
* Global assessment of functioning (DSM IV TR) less than 50
* Age less than 18 or greater than 60
* BMI lower than 18.5 or higher than 28
* Any history of Alcohol or substance dependence or abuse according to DSM-IV criteria (except for caffeine dependence)
* Any medical condition which in the opinion of the investigator may have an effect on mood symptoms
* Any individual who has a current mood disturbance (as defined by DSM-IV-R criteria)
* Use of cigarettes or other nicotine-containing products
* Allergy or other contraindication to uridine
* Individuals unable to comply with instructions or procedures of study
* History of significant head trauma
* Claustrophobia or other contraindication to MRI (e.g., pacemaker, metal fragments)
* Any illicit substance use in the past thirty days
* Any past treatment for substance abuse
* Any past hospitalization for mental illness.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Using MRI and MRS, after uridine administration an increase in brain GABA and NTP levels will be seen and increases in GABA and NTP will be correlated | after 7 days of treatment
  This choice of time period will allow a determination of time course to efficacy between the acute and extended ranges, and further, because therapeutic dosage levels of uridine have yet to be established, in this and future studies we hope to determine the optimal dosage at which uridine increases brain GABA and ß-NTP levels.

CONTACTS AND LOCATIONS:
Overall Officials: Perry F Renshaw, MD PhD, Principal Investigator — The Brain Institute, University of Utah
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States